CLINICAL TRIAL: NCT05422248
Title: Oxygen Wound Therapy Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIA-297
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Chronic Leg Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Series (Active Comparator): Standard wound care for 4 weeks followed by intervention device wound care for up to 12 weeks.
  Interventions: Device: Series Topical Oxygen Therapy
- Paired (Active Comparator): Intervention device wound care to a portion of wound and standard wound care to the remaining portion of the wound, for up to 12 weeks.
  Interventions: Device: Paired Topical Oxygen Therapy

INTERVENTIONS:
Device: Series Topical Oxygen Therapy — Standard care provided to the whole wound followed by intervention device care to the whole wound.
  Arms: Series
Device: Paired Topical Oxygen Therapy — Care provided to one portion of wound by intervention device and standard care to remaining portion of wound.
  Arms: Paired

SUMMARY:
Determine the feasibility of using a new topical oxygen therapy device to treat hard to heal lower leg wounds.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hard to heal lower leg wounds as determined by the treating clinician.
* Patient has a wound area greater than the area of the interface
* Aged 16 years and over
* Able to provide informed consent

Exclusion Criteria:

* Lower limb wounds with bone or tendon exposed
* Infected wounds which require treatment with antibiotics
* Wounds with critical bioburden requiring a medicated dressing
* Wounds that require dressing changes more than every second day, for example high exudating wounds
* Wounds with slough covering more than 30% of the wound surface

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in wound area | 12 weeks
  cm^2

CONTACTS AND LOCATIONS:
Overall Officials: Jolanta Krysa, Principal Investigator — Southern DHB Vascular Surgery
Locations (1):
- Otago Vascular Diagnostics, Dunedin, Otago, New Zealand